CLINICAL TRIAL: NCT01234571
Title: Impact of Hemo-dialysis Therapy on Blood Levels of Treprostenil in End Stage Renal Disease Patients With Pulmonary Hypertension
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dr. Mordechai Yigla, Rambam Health Care Campus
Other Study IDs: 0273-10CTIL
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-10

CONDITIONS: Pulmonary Hypertension; End-Stage Renal Disease; Hemo-dialysis Therapy
Keywords: Pulmonary hypertension; Remodulin (Treprostenil sodium); End-stage renal disease; Hemo-dialysis
MeSH Terms: conditions — Hypertension, Pulmonary; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Remodulin (Treprostenil sodium) is synthetic prostacyclin analog available as a solution for administration in the intravenous route. It is approved for treatment of class I - pulmonary hypertension functional capacity stage III-IV. A key factor for the success of pulmonary hypertension therapy is maintaining near constant blood level of a given medications along the day. A sudden decrease in the blood levels might lead to rebound phenomenon; abrupt increase in the pulmonary artery pressure which might lead to acute right ventricular failure and even to sudden death. As some PHT patients suffer are on hemo-dialysis therapy due to end-stage renal disease there is a need to document the variation of the blood level along the dialysis cycle.

DETAILED DESCRIPTION:
After giving informed consent 10 ml of blood will be drawn from the study population at the following occasions.

* Baseline measurement immediately before starting HD therapy.
* During the hemo-dialysis therapy - every one hour.
* After the end of the hemo-dialysis therapy - every one hour (a total of four measurements) to record recovery of Treprostenil blood levels.

ELIGIBILITY:
Inclusion Criteria:patients with PAH who receive chronic (more than 3 months) Treprostenil treatment administered intravenously as a single agent therapy who maintain chronic hemo-dialysis therapy. Patients must be in stable condition for at least one month. Patients other than class I PAH will be not included in this study.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with PAH who receive chronic (more than 3 months) Treprostenil treatment administered intravenously as a single agent therapy who maintain chronic hemo-dialysis therapy. Patients must be in stable condition for at least one month. Patients other than class I PAH will be not included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2010-11